CLINICAL TRIAL: NCT06416826
Title: An Investigation of the Effects of Rhythmic Sensory Stimulation on Fibromyalgia
Brief Title: Rhythmic Sensory Stimulation on Fibromyalgia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unforeseen circumstances
Sponsor: Women's College Hospital (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: FibroMusicTherapy
Record Dates: First submitted 2019-04-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain, Widespread
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): healthy controls
  n = 10
- patients (Active Comparator): patients with fibromyalgia
  n =20
  Interventions: Device: Vibroacoustic Therapy System - VTS 1000

INTERVENTIONS:
Device: Vibroacoustic Therapy System - VTS 1000 — Participants will undertake 15 self-administered sessions of RSS 40Hz low frequency sound stimulation, 30 minutes daily, over 3 weeks (5 days/week).
  Other Names: Rhythmic Sensory Stimulation
  Arms: patients

SUMMARY:
The aim of this project is to further examine the effectiveness of Rhythmic Sensory Stimulation (RSS) with low-frequency sounds and somatosensory stimulation as a complementary therapy for fibromyalgia, and to investigate potential mechanisms underlying the effects of RSS on chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical diagnosis of fibromyalgia
* able to read and write English adequately
* have satisfactory hearing bilaterally (self-reported)
* have the ability to operate the supplied device

Exclusion Criteria:

* acute and active inflammatory conditions (e.g., rheumatoid arthritis, osteoarthritis, autoimmune disease)
* medical or psychiatric illness
* history of psychosis, epilepsy, seizures
* pregnancy or breast feeding
* hemorrhaging or active bleeding
* thrombosis, angina pectoris
* heart disease, such as hypotension, arrhythmia, pacemaker
* substance abuse (harmful or hazardous use of psychoactive subtances, including alcohol and illicit drugs) in the last year
* suffering from a recently prolapsed vertebral disc
* recovering from a recent accident with back or neck injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
change in inflammatory cytokine levels | baseline, 1 month, 2 months
  The investigator will use a multiplex enzyme-linked immunosorbent assay (ELISA) to asses inflammatory cytokines in fibromyalgia.

SECONDARY OUTCOMES:
change in pain severity | baseline, 1 month, 2 months
  Patients will rate their pain severity on a scale from 0 (no pain) to 10 (extreme pain)
change in EEG brain activity | baseline, 1 month, 2 months
  The investigators will measure EEG dynamics to quantify dysfunctional activity in brain areas that are affected by fibromyalgia

IPD SHARING:
Plan to Share IPD: Undecided